CLINICAL TRIAL: NCT02911233
Title: Evaluation of Clot Stability Induced by Solulin: Evaluation of New Solulin Mutants Lacking Protein C Activation Capacity
Acronym: SOLUCLOT
Status: Completed | Type: Observational
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Other Study IDs: 13-136
Record Dates: First submitted 2016-09-07; First posted 2016-09-22 (Estimated); Last update posted 2016-09-22 (Estimated); Status verified 2016-09

CONDITIONS: Hemophilia A
MeSH Terms: conditions — Hemophilia A

STUDY DESIGN:
Time Perspective: Prospective

INTERVENTIONS:
Biological: Thromboelastograpgy

SUMMARY:
Hemophilia A is a rare X chromosome-linked recessive bleeding disorder that concerns one individual in 5000. In its severe form, hemophilia A is a life-threatening, crippling hemorrhagic disease. The treatment of bleeding episodes in hemophilia A patients involves the administration of exogenous human FVIII to restore normal hemostasis. The main complication of the substitutive treatment of hemophilia A is the development, in 15 to 30% of the cases, of anti-FVIII antibodies (FVIII inhibitors) that neutralize the pro-coagulant activity of therapeutically administered FVIII. In 2003, the average annual cost of care for a patient with hemophilia A was evaluated to be equal to 63,000 euros (2), which, in France (6000 patients), represents an annual budget of 378 million euros.

In order to reduce the cost of treatment and to bypass this complication, different therapeutic strategies (new products or adjunctive therapeutic options) have been explored, including platelet infusion, tranexamic acid, amino caproic acid, molecules that block tissue factor pathway inhibitor, combination of phospholipid -Factor Xa- Factor XIII and antibodies directed to the Tissue Factor Inhibitor Pathway (TFPI). Recently, Soluble thrombomodulin (Solulin) have been developed. This molecule may be used to partially correct the premature lysis defect in Factor VIII deficient plasma through an activated TAFI - dependent mechanism.

With a long half-life (15- to 30-hour) and effective dose range estimated to range from the sub-nanomolar to approximately 40nM, Solulin could potentially be administered on a weekly basis and provide the basis for a factor-sparing regime that would cut costs and make therapy more widely available. However, before proceeding to advanced trials, safety concerns stemming from the anticoagulant properties of Solulin must be addressed. The development of Solulin mutants lacking protein C activation capacity would make this concern redundant. At the same time, such mutant molecules are likely to possess an effective dose range.

Our project is to compare the behavior of recombinant Solulin and mutants of Solulin lacking protein C activation capacity with respect to their ability to stabilize fibrin clots in whole blood of humans with different coagulation factor deficiencies (hemophilia A, hemophilia B and rare blood coagulation deficiencies (factor X, VII, V).

ELIGIBILITY:
Inclusion Criteria:

* Patients with congenital blood disorder (hemophilia A and B),
* Inform consent

Exclusion Criteria:

* Patients with acquired blood disorder.
* Allo-immunisation against blood coagulation factor concentrates (FVIII inhibitor)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: - Patients with congenital blood disorder hemophilia A and B
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2014-03; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Evaluation of blood clot firmness in ROTEM experiments using mutant Solulin | 2 hours
Evaluation of fibrinolysis in ROTEM experiments using mutant Solulin | 2 hours

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital, Caen, Calvados, France